CLINICAL TRIAL: NCT06457594
Title: Prospective Cohort Analysis - the Role of General and Specific Patient Reported Outcome and Experience Measures Among Head and Neck Cancer Patients
Brief Title: Prospective PROM and PREM Analysis Demonstrating Specification Advantage and Language Barriers
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: QOL HMO-CTIL
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — EORTC QLQ-INFO25 EORTC QLQ - H&N43 and EORTC QLQ-C30

SUMMARY:
Importance:

Patient reported outcome and experience measures (PROM and PREM) constitute a cornerstone of the collective efforts to improve and personalize healthcare systems. The EORTC quality of life (QOL) group developed instruments evaluating general and disease specific oncology QOL questionnaires, and the quality of information received. Implementation of PREM and relevant PROM is essential for equity, better resources utility, accessibility and patient centered treatment.

Objectives:

The investigators describe the EORTC INFO 25 translation process followed by investigation of subpopulation where action is most needed. The investigators investigate which QOL questionnaire better reflects clinical parameters among head and neck cancer (HNC) patients.

Design:

A prospective cohort. Setting Tertiary, referral, head and neck dedicated surgical service.

Participants:

Consecutive head and neck cancer adult patients, surgically treated, recruited between January to December 2022.

Exposures:

The investigators prospectively analyzed the new EORTC INFO 25 Hebrew questionnaire together with previously established Arabic translated version and the general (QLQ-C30) and specific (QLQ - H&N43) oncology QOL questionnaires.

Main Outcomes and Measures:

Analyzing the quality of information provided and desired in diverse HNC subgroup of patients.

Analyzing which of PROM questionnaire better reflects HNC patients' disease and treatment parameters, which in turn, may predict poorer QOL.

Results:

The investigators recruited 60 patients, consisting of equal female: male ratio, of which 16.66% were native Arabic speaking. Validated INFO 25 scores (median 62.6±17.5) were not associated with patients' age, sex, education status, disease, and treatment parameters. Yet, the Arabic spoken sub-population had significantly lower scores (p<0.001).

In contrast to QLQ-C30, clinical imperative associations were demonstrated between QLQ - H&N43 and patients' disease stage (P<0.001), admission days (p<0.0001), free flap reconstruction (P<0.001) and adjuvant radiotherapy (P<0.001).

Conclusions and relevance:

The final version of the native EORTC INFO25 translation was approved by the EORTC. The investigators demonstrate lower INFO25 scores among the Arabic speaking population, suggesting frail equity and accessibility. In order to improve patients' centered treatment and resource utilization, the investigators reveal a strong association between disease severity and treatment aggressiveness and poor quality of life on specific, HNC oriented, EORTC QLQ - H&N43 questionnaire that was not validated on EORTC QLQ-C30, which can be omitted.

ELIGIBILITY:
Main inclusion Criteria:

* Adult patients (≥18 years)
* Head and Neck cancer patients surgically treated

Main exclusion Criteria:

* Illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive head and neck cancer patients were prospectively recruited between January to December 2022 at referral outpatient surgical clinics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Questionnaire scores | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No